CLINICAL TRIAL: NCT06744426
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 4-period, Crossover Phase I Study to Evaluate the Pharmacokinetics and the Safety After Administration of BR1015 and Co-administration of BR1015-3 and BR1015-2 in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and the Safety After Administration of BR1015 and Co-administration of BR1015-3 and BR1015-2 Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FIC-CT-103
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR1015 (Experimental)
  Interventions: Drug: BR1015
- BR1015-2 + BR1015-3 (Active Comparator)
  Interventions: Drug: BR1015-2; Drug: BR1015-3

INTERVENTIONS:
Drug: BR1015 — One tablet administered alone
  Arms: BR1015
Drug: BR1015-2 — One tablet administered alone
  Arms: BR1015-2 + BR1015-3
Drug: BR1015-3 — One tablet administered alone
  Arms: BR1015-2 + BR1015-3

SUMMARY:
The purpose of this clinical trial is to evaluate the pharmacokinetics and the safety after administration of BR1015 and co-administration of BR1015-3 and BR1015-2 in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Those weigh 50 kg or more and have body mass index (BMI) within the range of 18.0 to 30.0kg/m2 at screening visit.
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial*(Except for hormone drugs) from the date of consent to 14 days after the last administration and disagrees to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of non hormonal intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, contraceptive diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken drugs concerned about affecting this clinical trial within 10 days prior to the first day of administration. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 6 months prior to the first administration date.(However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrointestinal resection or gastrointestinal diseases that may affect the absorption of drugs. (Except for simple appendectomy, hernia surgery)
* Those who can't discontinue a diet (ex. raw grapefruit, grapefruit juice or food containing grapefruit, etc.) that may affect the absorption, distribution, metabolism, and excretion of the drug within 48 hours prior to the first day of administration.
* In the case of a female subject, those suspected pregnancy, pregnant woman, lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-04 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to time τ | 0-72 hours after administration
Maximum concentration of drug in plasma | 0-72 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No